CLINICAL TRIAL: NCT00956345
Title: A Multi-Centre, Multi-National, Open-Label, Dose Escalation Trial Evaluating Safety and Pharmacokinetics of Ascending Intravenous Doses of 40K Pegylated Recombinant FIX in Non-Bleeding Patients With Haemophilia B.
Brief Title: Safety of 40K Pegylated Recombinant Factor IX in Non-Bleeding Patients With Haemophilia B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-3639; 2009-011085-28 (EudraCT Number); 090857 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25U/kg (Experimental)
  Interventions: Drug: nonacog beta pegol
- 50U/kg (Experimental)
  Interventions: Drug: nonacog beta pegol
- 100U/kg (Experimental)
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — Cohort to receive a single dose of 25U/kg nonacog beta pegol administered intravenously (into the vein)
  Other Names: 40K PEG-rFIX
  Arms: 25U/kg
Drug: nonacog beta pegol — Cohort to receive a single dose of 50U/kg nonacog beta pegol administered intravenously (into the vein)
  Other Names: 40K PEG-rFIX
  Arms: 50U/kg
Drug: nonacog beta pegol — Cohort to receive a single dose of 100U/kg nonacog beta pegol administered intravenously (into the vein)
  Other Names: 40K PEG-rFIX
  Arms: 100U/kg

SUMMARY:
This trial is conducted in Europe, Japan and the United States of America (USA).

The aim of this clinical trial is to investigate the safety and pharmacokinetics (the determination of the concentration of the administered medication in blood over time) of Pegylated Recombinant Factor IX (nonacog beta pegol) in Non-Bleeding Patients with Haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with haemophilia B (baseline level of Factor IX less than or equal to 2%)
* History of at least 150 exposure days to any Factor IX products
* Body Mass Index (BMI) below 30.0 kg/m2 (inclusive)

Exclusion Criteria:

* History of Factor IX inhibitors
* Platelet count less than 50,000 platelets/microlitre (assessed by laboratory)
* Kidney or liver dysfunction
* Scheduled surgery requiring Factor IX replacement therapy, during the trial period

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs), Serious Adverse Events (SAEs) and Medical Events of Special Interests (MESIs) reported during the trial period | assessed up to five weeks after trial product administration
Antibody formation against 40K PEG-rFIX and test for inhibitors (Bethesda) | assessed up to five weeks after trial product administration

SECONDARY OUTCOMES:
AUC, CL, T½, Incremental recovery (first sample) from 0 to 48 hours after trial product administration | assessed up to five weeks after trial product administration
AUC, CL, T½, Incremental recovery (first sample) from 0 to 168 hours after trial product administration | assessed up to five weeks after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (18):
- United States (3):
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Novo Nordisk Investigational Site, Copenhagen, Denmark
- France (2):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lyon
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Hanover
- Japan (3):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Stockholm, Sweden
- United Kingdom (3):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Background] Negrier C, Knobe K, Tiede A, Giangrande P, Moss J. Enhanced pharmacokinetic properties of a glycoPEGylated recombinant factor IX: a first human dose trial in patients with hemophilia B. Blood. 2011 Sep 8;118(10):2695-701. doi: 10.1182/blood-2011-02-335596. Epub 2011 May 9. PMID 21555744
- [Background] Collins PW, Moss J, Knobe K, Groth A, Colberg T, Watson E. Population pharmacokinetic modeling for dose setting of nonacog beta pegol (N9-GP), a glycoPEGylated recombinant factor IX. J Thromb Haemost. 2012 Nov;10(11):2305-12. doi: 10.1111/jth.12000. PMID 22998153
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com